CLINICAL TRIAL: NCT01705067
Title: A Retro-Prospective, Non-randomized, Consecutive Series, SIngle Cohort, Multicenter Adaptive Design Study to Evaluate the Outcomes of Total Knee Arthroplasty (TKA) Using JOURNEY™ II BCS TotaL Knee SystEm (The NIMBLE Study)
Brief Title: Safety and Efficacy of the Journey II BCS Total Knee System
Acronym: NIMBLE
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011JBCK151
Record Dates: First submitted 2012-06-21; First posted 2012-10-12 (Estimated); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Degenerative Knee Disease; Total Knee Arthroplasty (TKA)
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Journey II BCS TKA: Subjects who previously received TKA with Journey II BCS Total Knee System
  Interventions: Device: TKA with Journey II BCS Total Knee System

INTERVENTIONS:
Device: TKA with Journey II BCS Total Knee System — TKA with Journey II BCS Total Knee System
  Other Names: Journey II BCS

SUMMARY:
Assess the safety and efficacy of the JOURNEY II BCS Total Knee System in subjects with degenerative knee disease requiring primary total knee replacement.

DETAILED DESCRIPTION:
Assess the safety and efficacy of the JOURNEY II BCS Total Knee System in subjects with degenerative knee disease requiring primary total knee replacement. Pre-operative and operative assessments collected retrospectively. All postoperative assessments beginning at the 6 month post-operative time point collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Subject received primary total knee arthroplasty with the JOURNEY™ II BCS Total Knee System due to degenerative joint disease
* Subject is willing to sign and date an IRB approved consent form
* Subject is of legal age to consent
* Subject plans to be available through ten (10) years postoperative follow-up
* Subject agrees to follow the study protocol

Exclusion Criteria:

* Subject received the JOURNEY™ II BCS Total Knee System on the affected knee as a revision for a previously failed total or unicondylar knee arthroplasty
* Subject received TKA on the contralateral knee as a revision for a previously failed total or unicondylar knee arthroplasty
* Subject possesses a contralateral or ipsilateral revision hip arthroplasty
* Subject has ipsilateral hip arthritis resulting in flexion contracture
* At the time of enrollment, subject has one or more of the following arthroplasties that are not fully healed and well-functioning, as determined by the investigator:

  * Ipsilateral or contralateral primary total hip arthroplasty or hip resurfacing arthroplasty
  * Contralateral primary total knee or unicondylar knee arthroplasty
* At the time of surgery, subject had an active infection or sepsis (treated or untreated)
* At the time of surgery, subject had presence of malignant tumor, metastatic, or neoplastic disease
* At the time of surgery, subject had conditions that may interfere with the TKA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease)
* At the time of surgery, subject had contralateral lower extremity condition causing abnormal ambulation
* Subject is pregnant or plans to become pregnant during the study
* Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study
* At the time of surgery, subject had a BMI>40
* At the time of enrollment, subject has a BMI>40
* Subject is enrolled in another investigational drug, biologic, or device study
* Subject is facing current or impending incarceration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects receiving the JOURNEY™ II BCS Total Knee System
Sampling Method: Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2012-06; Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of ITB Friction Pain | 6 months post-operatively

SECONDARY OUTCOMES:
Adverse Events | 6 months post-operatively, 1 year post-operatively, 2 years post-operatively, 5 years post-operatively, and 10 years post-operatively
Radiographic Evaluation | Baseline and 6 months post-operatively, 1 year post-operatively, 2 years post-operatively, 5 years post-operatively, and 10 years post-operatively
Knee Society Score | 6 months post-operatively, 1 year post-operatively, 2 years post-operatively, 5 years post-operatively, and 10 years post-operatively

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Joint Replacement Institute at St. Vincent Medical Center, Los Angeles, California
  - Fort Wayne Orthopedics, Fort Wayne, Indiana
  - Methodist Sports Medicine/The Orthopedic Specialist, Indianapolis, Indiana
  - Hospital for Special Surgery, New York, New York
  - OrthoCarolina, Charlotte, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Wellington Orthopaedics, Cincinnati, Ohio
  - Cincinnati Orthopaedic Research Institute, Cincinnati, Ohio
  - Minimally Invasive Orthopaedics, Columbus, Ohio
  - Tennessee Orthopaedic Clinics, Knoxville, Tennessee
  - San Antonio Orthopaedic Specialists, San Antonio, Texas
  - Evergreen Orthopaedic Clinic, Kirkland, Washington